CLINICAL TRIAL: NCT01168232
Title: A Phase II Evaluation of Ixabepilone (NSC #710428) in the Treatment of Recurrent or Persistent Carcinosarcoma of the Uterus
Brief Title: Ixabepilone in Treating Patients With Recurrent or Persistent Uterine Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02056; NCI-2011-02056 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0130F; CDR0000681684; GOG-0130F (Other: NRG Oncology); GOG-0130F (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Recurrent Uterine Corpus Sarcoma; Uterine Carcinosarcoma
MeSH Terms: interventions — ixabepilone; Epothilones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ixabepilone) (Experimental): Patients receive ixabepilone IV over 3 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixabepilone; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ixabepilone — Given IV
  Other Names: (1S,3S,7S,10R,11S,12S,16R)-7,11-Dihydroxy-8,8,10,12,16-pentamethyl-3-[(1E)-1-methyl-2-(2-methyl-4-thiazolyl)ethenyl]-17-oxa-4-azabicyclo[14.1.0]heptadecane-5,9-dione; Azaepothilone B; BMS 247550; BMS-247550; BMS247550; Epothilone; Epothilone-B BMS 247550; Ixempra
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and how well ixabepilone works in treating patients with persistent or recurrent uterine cancer. Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells of by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate of ixabepilone in patients with persistent or recurrent carcinosarcoma of the uterus.

II. To determine the nature and degree of toxicity of ixabepilone in this cohort of patients.

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free survival and overall survival.

TERTIARY OBJECTIVES:

I. To examine the expression of class III beta-tubulin in carcinosarcoma of the uterus.

II. To explore the association between class III beta-tubulin expression in carcinosarcoma of the uterus and response, progression-free and overall survival.

OUTLINE:

Patients receive ixabepilone IV over 3 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed uterine carcinosarcoma which is persistent or recurrent with documented disease progression after appropriate local therapy; acceptable histologic type is defined as carcinosarcoma (malignant mixed muellerian tumor), homologous or heterologous type
* All patients must have measurable disease; measurable disease is defined by Response Evaluation Criteria In Solid Tumors (RECIST) (version 1.1); measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one ?target lesion? to be used to assess response on this protocol as defined by RECIST version 1.1; tumors within a previously irradiated field will be designated as ?non-target? lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG Phase III or Rare Tumor protocol for the same patient population
* Patients must have a GOG Performance Status of 0, 1, or 2
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
  * Any other prior therapy directed at the malignant tumor, including biological and immunologic agents, must be discontinued at least three weeks prior to registration
* Patients must have had one prior chemotherapeutic regimen for management of carcinosarcoma; initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen
* Patients who have NOT received prior therapy with a taxane (such as paclitaxel or docetaxel) MUST receive a second regimen that includes a taxane
* Patients must have NOT received any additional cytotoxic chemotherapy except as noted above
* Patients are allowed to receive, but are not required to receive, one additional non-cytotoxic regimen for management of recurrent or persistent disease according to the following definition:

  * Non-cytotoxic (biologic or cytostatic) agents include (but are not limited to) monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
* Bilirubin less than or equal to 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Neuropathy (sensory and motor) less than or equal to grade 1
* Patients who have met the pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test 72 hours prior to the study entry and be practicing an effective form of contraception
* Patients who have received prior therapy with Ixabepilone
* Patients with a known history of severe (Common Terminology Criteria for Adverse Events [CTCAE] version [v]4.0) grade 3 or 4 hypersensitivity reaction to agents containing Cremophor? EL or its derivatives (eg, polyoxyethylated castor oil)
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, and other specific malignancies, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of uterine carcinosarcoma within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of uterine carcinosarcoma within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-09-07 (Actual); Primary Completion 2013-11-26 (Actual); Study Completion 2013-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn McCourt, Principal Investigator — NRG Oncology
Locations (78):
- United States (78):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - John Muir Medical Center-Concord Campus, Concord, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Florida Hospital Orlando, Orlando, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 9/7/2010 and closed to accrual on 8/26/2013 (suspended from 3/5/2012 to 9/30/2012).
Groups:
- Ixabepilone: Ixabepilone administered at 40 mg/m2 IV infusion over 3 hours on day 1 of a 21-day cycle until disease progression or adverse effects prohibit further treatment
Period: Overall Study
Arm/Group | Ixabepilone
Started | 42
Completed | 34 (Eligible and treated patients)
Not Completed | 8
Not completed — Ineligible-Second primary cancer site | 1
Not completed — Ineligible- Wrong cell type | 6
Not completed — Ineligible-Inadequate pathology | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Ixabepilone
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (7.7)
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0
  30-39 years | 0
  40-49 years | 0
  50-59 years | 7
  60-69 years | 13
  70-79 years | 12
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
International Federation of Gynecology and Obstetrics (FIGO) Stage - Recurrent/Persistent [Number; unit: participants] | 34
Histologic Type [Number; unit: participants]
  Carcinosarcoma-heterologus | 17
  Carcinosarcoma-homologous | 11
  Carcinosarcoma, MMT | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: Proportion of participants with objective tumor response. Objective tumor response is defined as complete or partial tumor response as assessed by RECIST 1.1.
Time Frame: Every other cycle for first 6 months; then every 3 months thereafter until completion of study treatment; and at any other time if clinically indicated based on symptoms or physical signs suggestive of progressive disease.1 cycle is 21 days
Population: Eligible and Treated Patients. Measure of dispersion is 95% One-sided confidence Interval
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Ixabepilone
Number analyzed (Participants) | 34
percentage | 11.8 [4.2 to 100]

2. Primary Outcome: Adverse Events (Grade 3 or Higher) During Treatment Period.
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v4.0
Time Frame: During treatment and up to 30 days after stopping the study treatment
Population: Eligible and Treated Participants
Measure: Number; unit: participants
Arm/Group | Ixabepilone
Number analyzed (Participants) | 34
participants
  Leukopenia | 15
  Thrombocytopenia | 0
  Neutropenia | 16
  Anemia | 5
  Other Investigations | 4
  Other Blood/lymphatics | 2
  Cardiac Disorders | 1
  Gastrointestinal disorders | 6
  General disorders and administration site conditio | 9
  Infections and infestations | 3
  Metabolism and nutrition disorders | 12
  Musculoskelatal and connective tissue disorders | 1
  Neoplasms benign, malignant and unspecified | 2
  Peripheral sensory neuropathy | 1
  Other nervous system disorders | 2
  Respitory, thoracic and mediastinal disorders | 5
  Vascular disorders | 8

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is the period of time from study entry to time of disease progression, death or date of last contact, whichever occurs first. Progression is assessed by RECIST 1.1
Time Frame: From study entry to disease progression, death or date of last contact, whichever occurs first, up to 5 years of follow-up.
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone
Number analyzed (Participants) | 34
months | 1.7 [1.3 to 4.2]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years of follow-up.
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone
Number analyzed (Participants) | 34
months | 7.7 [4.0 to 11.7]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during the patient's treatment and up to 30 days after stopping the study treatment are reported. The amount of time on study is specific to each patient.
Arm/Group | Ixabepilone
Serious Adverse Events (participants affected / at risk) | 17/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=34)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Death Nos (General disorders) | 1
Soft Tissue Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Lymphocyte Count Decreased (Investigations) | 2
Neutrophil Count Decreased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Neoplasms Benign, Malignant And Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=34)
Anemia (Blood and lymphatic system disorders) | 33
Sinus Bradycardia (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 2
Chest Pain - Cardiac (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Hearing Impaired (Ear and labyrinth disorders) | 4
Blurred Vision (Eye disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 12
Bloating (Gastrointestinal disorders) | 3
Rectal Mucositis (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 9
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 6
Oral Pain (Gastrointestinal disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 20
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Pain (General disorders) | 6
Neck Edema (General disorders) | 2
Malaise (General disorders) | 1
Localized Edema (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Edema Limbs (General disorders) | 4
Edema Face (General disorders) | 1
Fatigue (General disorders) | 24
Fever (General disorders) | 2
Chills (General disorders) | 1
Infusion Related Reaction (General disorders) | 1
Allergic Reaction (Immune system disorders) | 1
Skin Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Nail Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Weight Loss (Investigations) | 6
Weight Gain (Investigations) | 2
Platelet Count Decreased (Investigations) | 15
Lymphocyte Count Decreased (Investigations) | 4
Inr Increased (Investigations) | 1
Fibrinogen Decreased (Investigations) | 1
Creatinine Increased (Investigations) | 7
Neutrophil Count Decreased (Investigations) | 28
White Blood Cell Decreased (Investigations) | 29
Aspartate Aminotransferase Increased (Investigations) | 7
Alkaline Phosphatase Increased (Investigations) | 7
Alanine Aminotransferase Increased (Investigations) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 10
Hypercalcemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 12
Acidosis (Metabolism and nutrition disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 3
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tremor (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 19
Peripheral Motor Neuropathy (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Depressed Level Of Consciousness (Nervous system disorders) | 1
Concentration Impairment (Nervous system disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 3
Urinary Frequency (Renal and urinary disorders) | 4
Hematuria (Renal and urinary disorders) | 3
Vaginal Hemorrhage (Reproductive system and breast disorders) | 4
Pelvic Pain (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Nail Ridging (Skin and subcutaneous tissue disorders) | 1
Nail Loss (Skin and subcutaneous tissue disorders) | 2
Nail Discoloration (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 18
Thromboembolic Event (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less